CLINICAL TRIAL: NCT04059107
Title: Evaluation of 3D Printed Myoelectric Prosthetics in Children With Upper Congenital Limb Deficiency
Brief Title: Prosthetic Device in Children With Upper Congenital Limb Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Oregon Health and Science University (Other)
Collaborators: Limbitless Solutions (Unknown); University of Central Florida (Other)
Responsible Party: Principal Investigator, Albert Chi, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB17087
Record Dates: First submitted 2019-07-02; First posted 2019-08-16 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Upper Limb Deformities, Congenital
MeSH Terms: conditions — Upper Extremity Deformities, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prosthetic Device (Experimental): 3D Printed Myoelectric Prosthetic Device
  Interventions: Device: 3D Printed Myoelectric Prosthetic Device

INTERVENTIONS:
Device: 3D Printed Myoelectric Prosthetic Device — 3D Printed Myoelectric Prosthetic Device

SUMMARY:
This is a study being performed to evaluate the safety and effectiveness of 3D printed myoelectric prosthetic devices in children with a congenital upper limb deficiency.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about whether myoelectric prosthetic devices would be beneficial and useful for children. The study protocol specifies 4 study visits over the course of a year at the following intervals: baseline, 3 month, 6 month, 12 months. In following the protocol, each study visit will use the Assessment of Capacity for Myoelectric Control (ACMC) functional testing. The study participants will also complete several parent-child reported health related quality of life and musculoskeletal questionnaires. Specifically, the Pediatric Outcomes Data Collection Instrument (PODCI), the Pediatric Quality of Life Inventory (PedsQL), and the Children's Hand-Use Experience Questionnaire (CHEQ) will be used to measure efficacy of the myoelectric devices..

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 to 17 with congenital/infant upper limb deficiency identified by Limbitless Solutions will be referred to OHSU for evaluation and selection.
* All approved and consented subjects will receive a Limbitless 3D printed myoelectric device as delivered by established protocol.
* Preference will be given to children with long term previous experience with Limbitless Solutions' bionic systems.

Exclusion Criteria:

* Non English-speaking children and families. Due to the entirely volunteer nature of this project, the investigators are unable to hire appropriate translation services or create translated forms and surveys in other languages currently.
* Shoulder or wrist disarticulation will be excluded.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Measuring safety of the device through adverse event reporting. | 12 months
  The safety of the device will be measured through parental reporting and recorded observations of adverse events.
Children's experiences of using the myoelectric device while performing bi-manual tasks as assessed using a self-report questionnaire. | 12 months
  This assessment will measure the ability of the user to perform day-to-day tasks on three scales: grasp, performance time, and level of frustration.
Detects expected change in a person's ability to to do various functions while performing a specific task and scoring their motions. | 12 months
  This assessment will evaluate the ability of the myoelectric device use on functions that involve griping, holding, releasing, and coordinating between limbs using the Assessment of Capacity for Myoelectric Control (ACMC).
This self-report or parent-report tool is used to assess musculoskeletal health of the myoelectric device user. | 12 months
  This assessment contains six scales Upper Extremity Physical Function; Mobility/Transfers; Sports/Physical Function; Pain/Comfort; Happiness; and Global Function.
A self-report and parent-report sectional approach to measuring health-related quality of life. | 12 months
  This assessment uses four generic core scales including: physical health, emotional functioning, social functioning, and school functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Chi, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - The University of Central Florida, Orlando, Florida
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canfield MA, Honein MA, Yuskiv N, Xing J, Mai CT, Collins JS, Devine O, Petrini J, Ramadhani TA, Hobbs CA, Kirby RS. National estimates and race/ethnic-specific variation of selected birth defects in the United States, 1999-2001. Birth Defects Res A Clin Mol Teratol. 2006 Nov;76(11):747-56. doi: 10.1002/bdra.20294. PMID 17051527
- [Background] Blough DK, Hubbard S, McFarland LV, Smith DG, Gambel JM, Reiber GE. Prosthetic cost projections for servicemembers with major limb loss from Vietnam and OIF/OEF. J Rehabil Res Dev. 2010;47(4):387-402. doi: 10.1682/jrrd.2009.04.0037. PMID 20803406
- See also: Limbitless Solutions — http://limbitless-solutions.org/about-us/